CLINICAL TRIAL: NCT06359028
Title: An 8-Week, Randomized, Controlled, Examiner-Blind, Clinical Study to Evaluate the Efficacy of a Stannous Fluoride Toothpaste for the Relief of Dentin Hypersensitivity in a Population of Dentin Hypersensitivity Sufferers
Brief Title: Clinical Study to Evaluate the Anti-sensitivity Efficacy of a Stannous Fluoride Toothpaste in a Population of Dentin Hypersensitivity Sufferers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HALEON (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 300103
Record Dates: First submitted 2024-03-20; First posted 2024-04-11 (Actual); Results first posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Dentin Sensitivity
MeSH Terms: conditions — Dentin Sensitivity | interventions — hydrated silica gel-based toothpaste

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test toothpaste (Experimental): Participants will dose the toothbrush with a ribbon of toothpaste, across the full brush head and will brush the entire dentition thoroughly for at least 1-timed minute, twice daily (morning and evening), for approximately 56 days making sure to brush the sensitive areas of the two 'test teeth' carefully first. Participants who wish to rinse after brushing will be instructed to rinse with 10 milliliter (ml) water using graduated rinsing cup provided.
  Interventions: Drug: Stannous fluoride toothpaste
- Reference toothpaste (Negative control) (Active Comparator): Participants will dose the toothbrush with a ribbon of toothpaste, across the full brush head and will brush the entire dentition thoroughly for at least 1-timed minute, twice daily (morning and evening) for approximately 56 days. Participants who wish to rinse after brushing will be instructed to rinse with 10 ml water using graduated rinsing cup provided.
  Interventions: Drug: Crest cavity protection toothpaste

INTERVENTIONS:
Drug: Stannous fluoride toothpaste — Toothpaste containing 0.454 % weight/weight (w/w) SnF2
  Arms: Test toothpaste
Drug: Crest cavity protection toothpaste — Regular fluoride toothpaste containing 1100 parts per million (ppm) fluoride.
  Arms: Reference toothpaste (Negative control)

SUMMARY:
The aim of this study is to confirm the clinical Dentin Hypersensitivity (DH) efficacy of a 0.454 percent (%) Stannous Fluoride (SnF2) toothpaste.

DETAILED DESCRIPTION:
This will be a single center, 8-week, randomized, controlled, examiner-blind, 2-treatment arm, parallel design, stratified (by maximum baseline Schiff sensitivity score of the two selected 'test teeth') clinical study to evaluate the anti-sensitivity efficacy of a 0.454% SnF2 toothpaste in a DH population. The clinical efficacy of the 0.454% SnF2 toothpaste (test toothpaste) will be compared with that of a reference toothpaste, a commercially available, regular fluoride toothpaste with no known anti-sensitivity properties (negative control). Sufficient participants will be screened to randomize approximately 110 participants to investigational product (approximately 55 per treatment group) and to ensure approximately 100 evaluable participants complete the entire study (approximately 50 per treatment group).

ELIGIBILITY:
Inclusion Criteria:

* Participant provision of signed and dated informed consent before any study procedures are performed.
* Participant is male or female.
* Participant is 18 to 65 years of age, inclusive, at the time of signing the informed consent.
* Participant is willing and able to comply with the study visit schedule, product usage instructions, lifestyle restrictions and other study procedures.
* Participant is in good general, oral and mental health with, in the opinion of the investigator or medically qualified designee, no clinically significant or relevant abnormalities in self-reported medical history, or upon oral examination, that would impact their safety or wellbeing, or the outcomes of the study, if they were to participate in the study, or affect their ability to understand and follow study requirements.
* Screening (Visit 1): Participant must have-

  1. History of tooth sensitivity lasting more than six months but not more than 10 years (self-reported).
  2. Good general oral health, with a minimum of 20 natural teeth.
  3. Minimum of 2 accessible, non-adjacent teeth (incisors, canines, premolars), in different quadrants, which meet all of the following criteria:

     1. Exposed dentin due to facial/cervical erosion, abrasion or gingival recession (EAR).
     2. Modified Gingival Index (MGI) = 0 directly adjacent to the exposed dentin (that is, the test area only).
     3. Clinical mobility = 0
     4. Clinically confirmed DH to both tactile and evaporative (air) stimuli: a) Qualifying tactile threshold less than or equal to (<=) 20g. b) Qualifying Schiff sensitivity score more than or equal to (>=) 2.
* Baseline (Visit 2, Pre-Treatment)

  1. Participant must have a minimum of two, non-adjacent accessible teeth (incisors, canines, premolars), in different quadrants, with clinically confirmed DH to both tactile and evaporative (air) stimuli at both screening (Visit 1) and baseline (Visit 2).

     1. Qualifying tactile threshold <= 20g at screening and baseline.
     2. Qualifying Schiff sensitivity score >= 2 at screening and baseline.
  2. The clinical examiner will select two 'Test Teeth' from those which meet the tactile threshold and Schiff sensitivity score inclusion criteria at both screening and baseline. Notes: All teeth with clinically confirmed, qualifying levels of DH at screening (that is, a screening tactile threshold <= 20 g and a screening Schiff sensitivity score >= 2) will be assessed for tactile sensitivity at baseline. Teeth with a baseline tactile threshold <= 20g will then be assessed for baseline evaporative (air) sensitivity.

Exclusion Criteria:

* Participant is an employee of the investigator site directly involved in the conduct of the study, or an employee of the investigator site otherwise supervised by the investigator, or a member of their immediate family.
* Participant is an employee of the sponsor directly involved in the conduct of the study or a member of their immediate family.
* Female participant who is pregnant or intending to become pregnant during the study (self-reported).
* Female participant who is breastfeeding (self-reported).
* Participant with known or suspected intolerance or hypersensitivity to the study products, any of their stated ingredients or closely related compounds (self-reported).
* Participant with a recent history (within the last year) of alcohol or other substance abuse (self-reported).
* Participant is participating in or has participated in other studies (including non-medicinal studies) involving investigational product(s) within 30 days of screening (Visit 1) or plans to participate in other studies (including non-medicinal studies) during this study.
* Participant has participated in a tooth sensitivity study within 8 weeks of screening (Visit 1).
* Participant is currently using an oral care product indicated for DH relief or care of sensitive teeth or has used an anti-sensitivity product within 8 weeks of screening (Visit 1). Participants will be required to bring their current oral care products to screening (Visit 1) for staff to verify the absence of known anti-sensitivity ingredients and sensitivity-related claims on the product packaging/label text.
* Participant takes daily doses of medications/treatments which, in the opinion of the investigator or medically qualified designee, could interfere with their perception of tooth sensitivity (for example, analgesics, anticonvulsants, antihistamines that cause marked or moderate sedation, sedatives, tranquilizers, antidepressants, mood-altering and anti-inflammatory drugs).
* Screening (Visit 1): Participant has taken antibiotics in the 2 weeks prior to screening (Visit 1).
* Baseline (Visit 2, Pre-Treatment): Participant has taken antibiotics in the 2 weeks prior to baseline (Visit 2), that is, during the acclimatization period.
* Participant takes daily doses of a medication which, in the opinion of the investigator or medically qualified designee, is causing xerostomia.
* Participant requires antibiotic prophylaxis for dental procedures.
* Participant has had professional tooth de-sensitising treatment within 8 weeks of screening (Visit 1).
* Participant has had a tooth bleaching procedure within 8 weeks of screening (Visit 1).
* Participant has had dental prophylaxis within 4 weeks of screening (Visit 1).
* Participant has had treatment for periodontal disease (including surgery) within 12 months of screening (Visit 1).
* Participant has had scaling or root planning within 3 months of screening (Visit 1).
* Participant with gross periodontal disease.
* Participant with a tongue or lip piercing.
* Participant with evidence of gross intra-oral neglect or the need for extensive dental therapy.
* Participant with a fixed or removable partial prosthesis which, in the opinion of the investigator or dentally qualified designee, could impact study outcomes.
* Participant with multiple dental implants which, in the opinion of the investigator or dentally qualified designee, could impact study outcomes.
* Participant with fixed or removable orthodontic braces/bands or a fixed orthodontic retainer.
* Specific dentition exclusions for 'Test Teeth':

  1. Tooth with evidence of current/recent caries.
  2. Tooth with (self-reported) treatment for decay within 12 months of screening (Visit 1).
  3. Tooth with exposed dentin and deep, defective or facial restorations.
  4. Tooth with a full crown or veneer.
  5. Tooth adjacent to a bridge abutment or crown which, in the opinion of the investigator or dentally qualified designee, could impact study outcomes.
  6. Sensitive tooth with contributing etiologies other than EAR to exposed dentin.
  7. Sensitive tooth not expected to benefit from use of an anti-sensitivity toothpaste, in the opinion of the investigator or dentally qualified designee.
* Participant who, in the opinion of the investigator or designee, is unable to provide appropriate responses to the Labelled Magnitude Scale (LMS) training questions.
* Participant has previously been enrolled in this study.
* Participant who, in the opinion of the investigator or medically qualified designee, should not participate in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2024-03-25 (Actual); Primary Completion 2024-06-20 (Actual); Study Completion 2024-06-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Salus Research, Fort Wayne, Indiana, United States

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual participant data and study documents can be requested for further research from ww.clinical-trial-register@haleon.com
Supporting Information: Study Protocol, SAP, ICF
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months, but an extension can be granted, when justified, for up to another 12 months.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at a single center in the United States.
Pre-assignment Details: A total of 126 participants were screened into the study, 111 participants were enrolled, 104 participants were randomized to a treatment (53 participants in the test toothpaste group and 51 participants in the reference toothpaste group) and 102 participants completed the study (51 participants in the test toothpaste group and 51 participants in the reference toothpaste group).
Groups:
- Test Toothpaste: Participants were instructed to dose the toothbrush with a ribbon of test toothpaste, across the full brush head and to brush the entire dentition thoroughly for at least 1-timed minute, twice daily (morning and evening), for approximately 56 days making sure to brush the sensitive areas of the two 'test teeth' carefully first. Participants who wished to rinse after brushing were instructed to rinse with 10 milliliter (ml) water using the graduated rinsing cup provided.
- Reference Toothpaste (Negative Control): Participants were instructed to dose the toothbrush with a ribbon of reference toothpaste, across the full brush head and to brush the entire dentition thoroughly for at least 1-timed minute, twice daily (morning and evening) for approximately 56 days. Participants who wished to rinse after brushing were instructed to rinse with 10 ml water using the graduated rinsing cup provided.
Period: Overall Study
Arm/Group | Test Toothpaste | Reference Toothpaste (Negative Control)
Started | 53 | 51
Completed | 51 | 51
Not Completed | 2 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: The Safety population included all randomized participants who received at least one dose of investigational product.
Groups:
- Test Toothpaste: Participants were instructed to dose the toothbrush with a ribbon of test toothpaste, across the full brush head and to brush the entire dentition thoroughly for at least 1-timed minute, twice daily (morning and evening), for approximately 56 days making sure to brush the sensitive areas of the two 'test teeth' carefully first. Participants who wished to rinse after brushing were instructed to rinse with 10 ml water using the graduated rinsing cup provided.
- Total: Total of all reporting groups
Arm/Group | Test Toothpaste | Reference Toothpaste (Negative Control) | Total
Number analyzed (Participants) | 53 | 51 | 104
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.9 (8.27) | 49.9 (9.93) | 49.9 (9.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 43 | 92
  Male | 4 | 8 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 53 | 51 | 104
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American/African Heritage | 4 | 4 | 8
  American Indian or Alaskan Native | 1 | 0 | 1
  Asian - South East Asian Heritage | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  White - Arabic/North African Heritage | 0 | 2 | 2
  White - White/Caucasian/European Heritage | 46 | 44 | 90
  Multiple | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Adjusted Mean Change From Baseline in Schiff Sensitivity Score at Day 56
Description: Schiff sensitivity score was assessed by participant's response to an evaporative (air) stimulus after the stimulation of the 2 test teeth selected at Baseline by the examiner. Participant's response to the stimulus was evaluated by the examiner using the Schiff sensitivity scale immediately following administration of the evaporative air stimulus. Score ranged from 0-3, where 0=Does not respond to air stimulation; 1=Responds to air stimulus but does not request discontinuation of stimulus; 2=Responds to air stimulus and requests discontinuation or moves from stimulus; 3=Responds to stimulus, considers stimulus to be painful, requests discontinuation of the stimulus. Schiff sensitivity score = Mean score for the two 'Test Teeth' selected at baseline by the examiner. Change from baseline was calculated by subtracting baseline score from Day 56 score. A decrease in Schiff sensitivity score indicated an improvement.
Time Frame: Baseline and Day 56
Population: Modified Intent-To-Treat (mITT) population included all randomized participants who received at least one dose of investigational product and completed at least one-post Baseline dentin hypersensitivity (DH) efficacy assessment. Only those participants with data available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Test Toothpaste | Reference Toothpaste (Negative Control)
Number analyzed (Participants) | 51 | 51
score on a scale | -2.25 (0.080) | -0.31 (0.080)
Statistical Analysis 1: Comparison: Test Toothpaste vs Reference Toothpaste (Negative Control); Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures; Adjusted Mean Difference = -1.94, 95% CI 2-sided [-2.16 to -1.72], Standard Error of Mean 0.113

2. Secondary Outcome: Adjusted Mean Change From Baseline in Tactile Threshold at Day 56
Description: Tactile sensitivity was assessed by participant's response to tactile stimulus after the stimulation of the 2 test teeth selected at Baseline by the examiner. A constant pressure probe (Yeaple probe) was used for stimulation. The probe tip was placed perpendicular to the facial surface of tooth and drawn slowly across the exposed dentine. After each application, the participants were asked to indicate whether they experienced any pain or discomfort (yes/no response). The pressure setting with two consecutive 'yes' responses was recorded as the tactile threshold in gram (g). At baseline, the upper force setting was 20g. Tactile threshold (g) was derived as the mean value for the two 'Test Teeth' selected by the examiner at baseline. An increase in tactile threshold indicated an improvement in sensitivity. Change from baseline was calculated by subtracting baseline value from Day 56 value.
Time Frame: Baseline and Day 56
Population: mITT Population. Only those participants with data available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: gram
Arm/Group | Test Toothpaste | Reference Toothpaste (Negative Control)
Number analyzed (Participants) | 51 | 51
gram | 60.07 (2.539) | 2.70 (2.544)
Statistical Analysis 1: Comparison: Test Toothpaste vs Reference Toothpaste (Negative Control); Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures; Adjusted Mean Difference = 57.37, 95% CI 2-sided [50.23 to 64.51], Standard Error of Mean 3.599

3. Secondary Outcome: Adjusted Mean Change From Baseline in Schiff Sensitivity Score at Day 28
Description: Schiff sensitivity score was assessed by participant's response to an evaporative (air) stimulus after the stimulation of the 2 test teeth selected at Baseline by the examiner. Participant's response to the stimulus was evaluated by the examiner using the Schiff sensitivity scale immediately following administration of the evaporative air stimulus. Score ranged from 0-3, where 0=Does not respond to air stimulation; 1=Responds to air stimulus but does not request discontinuation of stimulus; 2=Responds to air stimulus and requests discontinuation or moves from stimulus; 3=Responds to stimulus, considers stimulus to be painful, requests discontinuation of the stimulus. Schiff sensitivity score = Mean score for the two 'Test Teeth' selected at baseline by the examiner. Change from baseline was calculated by subtracting baseline score from Day 28 score. A decrease in Schiff sensitivity score indicated an improvement.
Time Frame: Baseline and Day 28
Population: mITT Population.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Test Toothpaste | Reference Toothpaste (Negative Control)
Number analyzed (Participants) | 52 | 51
score on a scale | -1.75 (0.085) | -0.10 (0.086)
Statistical Analysis 1: Comparison: Test Toothpaste vs Reference Toothpaste (Negative Control); Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures; Adjusted Mean Difference = -1.65, 95% CI 2-sided [-1.89 to -1.41], Standard Error of Mean 0.121

4. Secondary Outcome: Adjusted Mean Change From Baseline in Tactile Threshold at Day 28
Description: Tactile sensitivity was assessed by participant's response to tactile stimulus after the stimulation of the 2 test teeth selected at Baseline by the examiner. A constant pressure probe (Yeaple probe) was used for stimulation. The probe tip was placed perpendicular to the facial surface of tooth and drawn slowly across the exposed dentine. After each application, the participants were asked to indicate whether they experienced any pain or discomfort (yes/no response). The pressure setting with two consecutive 'yes' responses was recorded as the tactile threshold in gram. At baseline, the upper force setting was 20g. Tactile threshold (g) was derived as the mean value for the two 'Test Teeth' selected by the examiner at baseline. An increase in tactile threshold indicated an improvement in sensitivity. Change from baseline was calculated by subtracting baseline value from Day 28 value.
Time Frame: Baseline and Day 28
Population: mITT Population.
Measure: Least Squares Mean (Standard Error); unit: gram
Arm/Group | Test Toothpaste | Reference Toothpaste (Negative Control)
Number analyzed (Participants) | 52 | 51
gram | 36.59 (3.009) | 1.23 (3.038)
Statistical Analysis 1: Comparison: Test Toothpaste vs Reference Toothpaste (Negative Control); Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures; Adjusted Mean Difference = 35.37, 95% CI 2-sided [26.88 to 43.86], Standard Error of Mean 4.280

5. Secondary Outcome: Adjusted Mean Change From Baseline in Impact on Everyday Life (Section 1 of Dentin Hypersensitivity Experience Questionnaire [DHEQ-48], Question [Q]7-9) at Days 28 and 56
Description: DHEQ section 1, questions 7-9 were about teeth sensation and its impact on everyday life. Participants scored Q7 (how intense are the sensations?) on a scale of 1 (not at all intense) to 10 (worst imaginable); Q8 (how bothered are you by any sensations?) on a scale of 1 (not at all bothered) to 10 (extremely bothered); Q9 (how well can you tolerate sensations?) on a scale of 1 (can easily tolerate) to 10 (can't tolerate at all). Thus, the total score ranged from 3 to 30; where the lower score indicated less sensitivity and less impact on everyday life. Change from baseline was calculated as score at indicated post-baseline timepoints minus score at baseline.
Time Frame: Baseline, Day 28 and Day 56
Population: mITT Population. Only those participants with data available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Test Toothpaste | Reference Toothpaste (Negative Control)
Number analyzed (Participants) | 52 | 51
score on a scale
  Q7, Day 28 | -1.44 (0.216) | -0.61 (0.199)
  Q7, Day 56: number analyzed (Participants) | 51 | 51
  Q7, Day 56 | -2.83 (0.217) | -0.71 (0.225)
  Q8, Day 28 | -1.69 (0.224) | -0.53 (0.216)
  Q8, Day 56: number analyzed (Participants) | 51 | 51
  Q8, Day 56 | -3.04 (0.222) | -0.78 (0.226)
  Q9, Day 28 | -0.46 (0.260) | -0.12 (0.216)
  Q9, Day 56: number analyzed (Participants) | 51 | 51
  Q9, Day 56 | -1.96 (0.260) | -0.43 (0.269)
Statistical Analysis 1: Comparison: Test Toothpaste vs Reference Toothpaste (Negative Control); Q7, Day 28; Test type: Superiority; p = 0.1268, Mixed Model with Repeated Measures; Adjusted Mean Difference = -0.46, 95% CI 2-sided [-1.04 to 0.13], Standard Error of Mean 0.296
Statistical Analysis 2: Comparison: Test Toothpaste vs Reference Toothpaste (Negative Control); Q7, Day 56; Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures; Adjusted Mean Difference = -1.75, 95% CI 2-sided [-2.38 to -1.13], Standard Error of Mean 0.316
Statistical Analysis 3: Comparison: Test Toothpaste vs Reference Toothpaste (Negative Control); Q8, Day 28; Test type: Superiority; p = 0.0245, Mixed Model with Repeated Measures; Adjusted Mean Difference = -0.72, 95% CI 2-sided [-1.35 to -0.09], Standard Error of Mean 0.315
Statistical Analysis 4: Comparison: Test Toothpaste vs Reference Toothpaste (Negative Control); Q8, Day 56; Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures; Adjusted Mean Difference = -1.81, 95% CI 2-sided [-2.44 to -1.18], Standard Error of Mean 0.318
Statistical Analysis 5: Comparison: Test Toothpaste vs Reference Toothpaste (Negative Control); Q9, Day 28; Test type: Superiority; p = 0.3851, Mixed Model with Repeated Measures; Adjusted Mean Difference = -0.29, 95% CI 2-sided [-0.96 to 0.37], Standard Error of Mean 0.337
Statistical Analysis 6: Comparison: Test Toothpaste vs Reference Toothpaste (Negative Control); Q9, Day 56; Test type: Superiority; p = 0.0002, Mixed Model with Repeated Measures; Adjusted Mean Difference = -1.48, 95% CI 2-sided [-2.22 to -0.73], Standard Error of Mean 0.375

6. Secondary Outcome: Adjusted Mean Change From Baseline in DHEQ Total Score (Section 2, Q1-34) at Days 28 and 56
Description: The DHEQ was a condition-specific measure of Oral Health-related Quality of Life (OHrQoL) in relation to DH which consisted of a total of 34 questions in section 2 grouped into 5 separate domains: Restrictions(Q1-4), Adaptation(Q5-16), Social Impact(Q17-21), Emotional Impact(Q22-29), and Identity(Q30-34), each scored using a 7-point scale ranging from 1 (strongly disagree) to 7 (strongly agree). Thus, the total score ranged from 34 to 238; where the lower score indicated improvement in the symptoms. Change from baseline was calculated as score at indicated post-baseline timepoints minus score at baseline.
Time Frame: Baseline, Day 28 and Day 56
Population: mITT Population. Only those participants with data available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Test Toothpaste | Reference Toothpaste (Negative Control)
Number analyzed (Participants) | 52 | 51
score on a scale
  Day 28 | -14.79 (3.833) | -7.47 (2.678)
  Day 56: number analyzed (Participants) | 51 | 51
  Day 56 | -34.56 (5.296) | -8.94 (3.394)
Statistical Analysis 1: Comparison: Test Toothpaste vs Reference Toothpaste (Negative Control); Day 28; Test type: Superiority; p = 0.1884, Mixed Model with Repeated Measures; Adjusted Mean Difference = -6.19, 95% CI 2-sided [-15.46 to 3.08], Standard Error of Mean 4.674
Statistical Analysis 2: Comparison: Test Toothpaste vs Reference Toothpaste (Negative Control); Day 56; Test type: Superiority; p = 0.0002, Mixed Model with Repeated Measures; Adjusted Mean Difference = -24.49, 95% CI 2-sided [-37.00 to -11.97], Standard Error of Mean 6.308

7. Secondary Outcome: Adjusted Mean Change From Baseline in DHEQ Restrictions Domain (Section 2, Q1-4) Score at Days 28 and 56
Description: Restrictions domain in DHEQ evaluated the ways in which any sensations in teeth affected participant's daily life. This consisted of 4 questions each scored using a 7-point scale ranging from 1 (strongly disagree) to 7 (strongly agree). Thus, the total score ranged from 4 to 28; where the lower score indicated improvement in the symptoms. Change from baseline was calculated as score at indicated post-baseline timepoints minus score at baseline.
Time Frame: Baseline, Day 28 and Day 56
Population: mITT Population. Only those participants with data available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Test Toothpaste | Reference Toothpaste (Negative Control)
Number analyzed (Participants) | 52 | 51
score on a scale
  Day 28 | -2.27 (0.634) | -1.20 (0.444)
  Day 56: number analyzed (Participants) | 51 | 51
  Day 56 | -4.94 (0.742) | -1.90 (0.492)
Statistical Analysis 1: Comparison: Test Toothpaste vs Reference Toothpaste (Negative Control); Day 28; Test type: Superiority; p = 0.3003, Mixed Model with Repeated Measures; Adjusted Mean Difference = -0.81, 95% CI 2-sided [-2.34 to 0.73], Standard Error of Mean 0.774
Statistical Analysis 2: Comparison: Test Toothpaste vs Reference Toothpaste (Negative Control); Day 56; Test type: Superiority; p = 0.0028, Mixed Model with Repeated Measures; Adjusted Mean Difference = -2.77, 95% CI 2-sided [-4.56 to -0.97], Standard Error of Mean 0.903

8. Secondary Outcome: Adjusted Mean Change From Baseline in DHEQ Adaptation Domain Score (Section 2, Q5-16) at Days 28 and 56
Description: Adaptation domain in DHEQ evaluated 'the ways in which the sensations in teeth have forced participants to change things in their daily life'; 'things they do in their daily life to avoid experiencing the sensations in their teeth'. This consisted of 12 questions each scored using a 7-point scale ranging from 1 (strongly disagree) to 7 (strongly agree). Thus, the total score ranged from 12 to 84; where the lower score indicated improvement in the symptoms. Change from baseline was calculated as score at indicated post-baseline timepoints minus score at baseline.
Time Frame: Baseline, Day 28 and Day 56
Population: mITT Population. Only those participants with data available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Test Toothpaste | Reference Toothpaste (Negative Control)
Number analyzed (Participants) | 52 | 51
score on a scale
  Day 28 | -6.45 (1.600) | -1.73 (1.396)
  Day 56: number analyzed (Participants) | 51 | 51
  Day 56 | -12.42 (2.530) | -3.31 (1.726)
Statistical Analysis 1: Comparison: Test Toothpaste vs Reference Toothpaste (Negative Control); Day 28; Test type: Superiority; p = 0.0784, Mixed Model with Repeated Measures; Adjusted Mean Difference = -3.78, 95% CI 2-sided [-8.00 to 0.44], Standard Error of Mean 2.127
Statistical Analysis 2: Comparison: Test Toothpaste vs Reference Toothpaste (Negative Control); Day 56; Test type: Superiority; p = 0.0092, Mixed Model with Repeated Measures; Adjusted Mean Difference = -8.17, 95% CI 2-sided [-14.27 to -2.07], Standard Error of Mean 3.074

9. Secondary Outcome: Adjusted Mean Change From Baseline in DHEQ Social Impact Domain (Section 2, Q17-21) Score at Days 28 and 56
Description: Social Impact domain in DHEQ evaluated the way the sensations affected participants when they were with other people or in certain situations. This consisted of 5 questions each scored using a 7-point scale ranging from 1 (strongly disagree) to 7 (strongly agree). Thus, the total score ranged from 5 to 35; where the lower score indicated improvement in the symptoms. Change from baseline was calculated as score at indicated post-baseline timepoints minus score at baseline.
Time Frame: Baseline, Day 28 and Day 56
Population: mITT Population. Only those participants with data available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Test Toothpaste | Reference Toothpaste (Negative Control)
Number analyzed (Participants) | 52 | 51
score on a scale
  Day 28 | -1.23 (0.644) | -0.94 (0.552)
  Day 56: number analyzed (Participants) | 51 | 51
  Day 56 | -3.63 (0.771) | -0.24 (0.587)
Statistical Analysis 1: Comparison: Test Toothpaste vs Reference Toothpaste (Negative Control); Day 28; Test type: Superiority; p = 0.8686, Mixed Model with Repeated Measures; Adjusted Mean Difference = -0.14, 95% CI 2-sided [-1.82 to 1.54], Standard Error of Mean 0.846
Statistical Analysis 2: Comparison: Test Toothpaste vs Reference Toothpaste (Negative Control); Day 56; Test type: Superiority; p = 0.0012, Mixed Model with Repeated Measures; Adjusted Mean Difference = -3.24, 95% CI 2-sided [-5.18 to -1.31], Standard Error of Mean 0.976

10. Secondary Outcome: Adjusted Mean Change From Baseline in DHEQ Emotional Impact Domain (Section 2, Q22-29) Score at Days 28 and 56
Description: Emotional Impact Domain in DHEQ evaluated the way the sensations in participant's teeth made them feel. This consisted of 8 questions each scored using a 7-point scale ranging from 1 (strongly disagree) to 7 (strongly agree). Thus, the total score ranged from 8 to 56; where the lower score indicated improvement in the symptoms. Change from baseline was calculated as score at indicated post-baseline timepoints minus score at baseline.
Time Frame: Baseline, Day 28 and Day 56
Population: mITT Population. Only those participants with data available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Test Toothpaste | Reference Toothpaste (Negative Control)
Number analyzed (Participants) | 52 | 51
score on a scale
  Day 28 | -4.10 (1.089) | -3.33 (0.957)
  Day 56: number analyzed (Participants) | 51 | 51
  Day 56 | -10.23 (1.340) | -2.98 (0.958)
Statistical Analysis 1: Comparison: Test Toothpaste vs Reference Toothpaste (Negative Control); Day 28; Test type: Superiority; p = 0.9047, Mixed Model with Repeated Measures; Adjusted Mean Difference = -0.17, 95% CI 2-sided [-3.04 to 2.69], Standard Error of Mean 1.444
Statistical Analysis 2: Comparison: Test Toothpaste vs Reference Toothpaste (Negative Control); Day 56; Test type: Superiority; p = 0.0001, Mixed Model with Repeated Measures; Adjusted Mean Difference = -6.66, 95% CI 2-sided [-9.95 to -3.38], Standard Error of Mean 1.656

11. Secondary Outcome: Adjusted Mean Change From Baseline in DHEQ Identity Domain (Section 2, Q30-34) Score at Days 28 and 56
Description: Identity Domain in DHEQ evaluated what the sensations in participant's teeth meant for them. This consisted of 5 questions each scored using a 7-point scale ranging from 1 (strongly disagree) to 7 (strongly agree). Thus, the total score ranged from 5 to 35; where the lower score indicated improvement in the symptoms. Change from baseline was calculated as score at indicated post-baseline timepoints minus score at baseline.
Time Frame: Baseline, Day 28 and Day 56
Population: mITT Population. Only those participants with data available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Test Toothpaste | Reference Toothpaste (Negative Control)
Number analyzed (Participants) | 52 | 51
score on a scale
  Day 28 | -0.69 (0.666) | -0.27 (0.517)
  Day 56: number analyzed (Participants) | 51 | 51
  Day 56 | -3.34 (0.735) | -0.51 (0.725)
Statistical Analysis 1: Comparison: Test Toothpaste vs Reference Toothpaste (Negative Control); Day 28; Test type: Superiority; p = 0.5733, Mixed Model with Repeated Measures; Adjusted Mean Difference = -0.47, 95% CI 2-sided [-2.14 to 1.19], Standard Error of Mean 0.840
Statistical Analysis 2: Comparison: Test Toothpaste vs Reference Toothpaste (Negative Control); Day 56; Test type: Superiority; p = 0.0060, Mixed Model with Repeated Measures; Adjusted Mean Difference = -2.88, 95% CI 2-sided [-4.92 to -0.84], Standard Error of Mean 1.026

12. Secondary Outcome: Adjusted Mean Change From Baseline in Global Oral Health (DHEQ Section 2, Q35) Score at Days 28 and 56
Description: Global Oral Health was evaluated using a single question which asked about the overall health of participant's mouth, teeth, and gums. The scale ranged from 1 (excellent) to 6 (Very poor), where the lower score indicated improvement in the symptoms. Change from baseline was calculated as score at indicated post-baseline timepoints minus score at baseline.
Time Frame: Baseline, Day 28 and Day 56
Population: mITT Population. Only those participants with data available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Test Toothpaste | Reference Toothpaste (Negative Control)
Number analyzed (Participants) | 52 | 51
score on a scale
  Day 28 | -0.15 (0.076) | -0.10 (0.100)
  Day 56: number analyzed (Participants) | 51 | 51
  Day 56 | -0.23 (0.082) | -0.06 (0.074)
Statistical Analysis 1: Comparison: Test Toothpaste vs Reference Toothpaste (Negative Control); Day 28; Test type: Superiority; p = 0.2768, Mixed Model with Repeated Measures; Adjusted Mean Difference = -0.14, 95% CI 2-sided [-0.39 to 0.11], Standard Error of Mean 0.127
Statistical Analysis 2: Comparison: Test Toothpaste vs Reference Toothpaste (Negative Control); Day 56; Test type: Superiority; p = 0.0232, Mixed Model with Repeated Measures; Adjusted Mean Difference = -0.26, 95% CI 2-sided [-0.48 to -0.04], Standard Error of Mean 0.113

13. Secondary Outcome: Adjusted Mean Change From Baseline in Effect on Life Overall (DHEQ Section 2, Q36-39) Score at Days 28 and 56
Description: Effect on life was evaluated using 4 questions which asked how much the sensations in teeth affected participant's life overall. The scale ranged from 0 (not at all) to 4 (Very much) and thus, the total score ranged from 0 to 16; where the lower score indicated improvement in the symptoms. Change from baseline was calculated as score at indicated post-baseline timepoint minus score at baseline.
Time Frame: Baseline, Day 28 and Day 56
Population: mITT Population. Only those participants with data available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Test Toothpaste | Reference Toothpaste (Negative Control)
Number analyzed (Participants) | 52 | 51
score on a scale
  Day 28 | -0.80 (0.253) | -0.53 (0.311)
  Day 56: number analyzed (Participants) | 51 | 51
  Day 56 | -1.93 (0.277) | -0.71 (0.261)
Statistical Analysis 1: Comparison: Test Toothpaste vs Reference Toothpaste (Negative Control); Day 28; Test type: Superiority; p = 0.8996, Mixed Model with Repeated Measures; Adjusted Mean Difference = 0.05, 95% CI 2-sided [-0.75 to 0.85], Standard Error of Mean 0.403
Statistical Analysis 2: Comparison: Test Toothpaste vs Reference Toothpaste (Negative Control); Day 56; Test type: Superiority; p = 0.0204, Mixed Model with Repeated Measures; Adjusted Mean Difference = -0.90, 95% CI 2-sided [-1.66 to -0.14], Standard Error of Mean 0.383

ADVERSE EVENTS:
Time Frame: From signing of informed consent form until 5 days after the last administration of study product or the last study procedure (up to approximately 90 days).
Description: An adverse event (AE) was defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study product including an acclimatization product (or medical device), whether or not considered related to the study product, including an acclimatization product (or medical device). A serious adverse event (SAE) is a particular category of AE where the adverse outcome is serious.
Arm/Group | Test Toothpaste | Reference Toothpaste (Negative Control)
All-Cause Mortality (participants affected / at risk) | 0/53 | 0/51
Serious Adverse Events (participants affected / at risk) | 0/53 | 0/51
Other Adverse Events (participants affected / at risk) | 5/53 | 4/51
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Test Toothpaste (N=53) | Reference Toothpaste (Negative Control) (N=51)
APHTHOUS ULCER (Gastrointestinal disorders) | 1 | 3
HYPERAESTHESIA TEETH (Gastrointestinal disorders) | 1 | 1
GLOSSODYNIA (Gastrointestinal disorders) | 1 | 0
LIP SWELLING (Gastrointestinal disorders) | 1 | 0
ORAL DISORDER (Gastrointestinal disorders) | 1 | 0
ORAL MUCOSAL EXFOLIATION (Gastrointestinal disorders) | 1 | 0
DEHYDRATION (Metabolism and nutrition disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
HALEON agreements may vary with individual investigators but will not prohibit any investigator from publishing. HALEON supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2024-02-06): https://cdn.clinicaltrials.gov/large-docs/28/NCT06359028/Prot_000.pdf
  • Statistical Analysis Plan (2024-05-03): https://cdn.clinicaltrials.gov/large-docs/28/NCT06359028/SAP_001.pdf